CLINICAL TRIAL: NCT03594955
Title: An Open-label, First-in-human, Dose Escalation Study of SAR440234 Administered as Single Agent by Intravenous Infusion in Patients With Relapsed or Refractory Acute Myeloid Leukemia (R/R AML), B-cell Acute Lymphoblastic Leukemia (B-ALL), or High Risk Myelodysplasia (HR-MDS)
Brief Title: First in Human Testing of Dose-escalation of SAR440234 in Patients With Acute Myeloid Leukemia, Acute Lymphoid Leukemia and Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED15138; 2017-004148-39 (EudraCT Number); U1111-1197-8041 (Other: UTN)
Record Dates: First submitted 2018-07-02; First posted 2018-07-20 (Actual); Results first posted 2022-04-07 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Leukaemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SAR440234 (Experimental): SAR440234 was administered as intravenous infusion once weekly for 6 weeks per Cycle. Per plan, participants were to receive first 2 to 3 doses as Lead-in doses followed by a fixed dose until the end of treatment or unless the dose needs to be decreased for safety reasons. Due to early study termination, all participants received only 1 treatment cycle at a dose of 1 nanogram per kilogram (ng/kg) once weekly.
  Interventions: Drug: SAR440234

INTERVENTIONS:
Drug: SAR440234 — Pharmaceutical form:lyophilisate to be resuspended in solution Route of administration: intravenous

SUMMARY:
Primary Objective:

* Dose escalation: To determine the maximum tolerated dose (MTD) of SAR440234 administered as a single agent in participants with relapsed or refractory acute myeloid leukemia (R/R AML), high risk myelodysplastic syndrome (HR-MDS), or B-cell acute lymphoblastic leukemia (B-ALL), and determine the recommended phase 2 dose (RP2D) for the subsequent Expansion part.
* Expansion part: To assess the activity of single agent SAR440234 at the RP2D in participants with R/R AML or HR-MDS.

Secondary Objective:

* To characterize the safety profile including cumulative adverse drug reactions.
* To evaluate the potential immunogenicity of SAR440234.
* To assess any preliminary evidence of hematologic response in the Dose Escalation Part.

DETAILED DESCRIPTION:
The duration of the study for the participants included a period for screening of up to 14 days. The cycle duration was 42 days. Participants continued study treatment as long as clinical benefit was possible or until disease progression, unacceptable adverse reaction, participant's decision to stop treatment, or other reason of discontinuation. After study treatment discontinuation participants returned to the study site 30 days after the last administration of SAR440234 for end of treatment assessments. Participants without documented disease progression at the end of a treatment visit who had not yet started treatment with another anti-cancer therapy would proceed with monthly follow-up visits until initiation of another anti-cancer therapy, disease progression, or study cut-off date, whichever came first.

ELIGIBILITY:
Inclusion criteria:

* Confirmed diagnosis of Acute Myeloblastic leukemia (AML) (except acute promyelocytic leukemia), or myelodysplastic syndrome (MDS) with a risk category of intermediate or higher. Participants must had exhausted available treatment options and might not be eligible for any treatment known to provide clinical benefit.
* Participants with AML must had relapsed or refractory disease that had been resistant to available therapies.
* Participants with B-ALL (B acute lymphoid leukemia) in second or subsequent relapse: should had completed previously greater than or equal to (>=) 1 cycle of a salvage regimen. Participants must had exhausted available treatment options and must not be eligible for any treatment known to provide clinical benefit.
* Participants with HR-MDS (high risk myelodysplastic syndrome) must have greater than (>) 10 percentage blasts in the bone marrow at the time of enrollment and fit one of the following categories: Not eligible for induction therapy and having completed >=2 cycles of therapy or not eligible for allogeneic stem cell transplant and had completed >=1 course of induction therapy.
* Signed written informed consent.

Exclusion criteria:

* Aged less than 16 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status >2.
* Participants with inadequate biological tests.
* White blood cell count > 30,000 per cubic millimeter.
* History of active or chronic autoimmune conditions that had required or requires therapy.
* Graft-versus-host disease following allogeneic stem cell transplantation required treatment with more than 10 milligrams (mg) of oral prednisone or equivalent daily. The stem cell transplant and/or donor lymphocyte infusion should had been performed more than 3 months before study treatment start.
* Second primary malignancy that required active therapy. Adjuvant hormonal therapy was allowed.
* Previous treatment with radiotherapy or immunotherapeutic agents in the 4 weeks prior to investigational medicinal product (IMP) administration.
* Previous treatment with any other investigational agent in the 4 weeks prior to IMP administration.
* Receiving, at the time of first IMP administration, of concurrent steroids >10 mg per day of oral prednisone or the equivalent for >=3 months.
* Requirement for tocilizumab for any other diagnosis.
* Evidence of active central nervous system leukemia at the time of enrollment.
* Acquired immunodeficiency syndrome (AIDS-related illnesses) or human immunodeficiency virus disease requiring antiretroviral treatment or had active Hepatitis B viral infection or Hepatitis C viral infection.
* Women of childbearing potential, male with a partner of childbearing potential who did not agree to use effective methods of birth control.
* Any clinically significant, uncontrolled medical conditions that, in the Investigator's opinion, would expose excessive risk to the participant or may interfere with compliance or interpretation of the study results.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2021-02-06 (Actual); Study Completion 2021-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- Investigational Site Number 8400001, Houston, Texas, United States
- France (3):
  - Investigational Site Number 2500004, Marseille
  - Investigational Site Number 2500001, Paris
  - Investigational Site Number 2500003, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Gerard E, Zohar S, Thai HT, Lorenzato C, Riviere MK, Ursino M. Bayesian dose regimen assessment in early phase oncology incorporating pharmacokinetics and pharmacodynamics. Biometrics. 2022 Mar;78(1):300-312. doi: 10.1111/biom.13433. Epub 2021 Feb 18. PMID 33527351

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 4 sites in France and the United States. A total of 12 participants were screened, of whom 5 participants were screen failures, mainly due to not meeting inclusion criteria. A total of 7 participants were enrolled and treated in Dose Escalation Part before termination of study.
Pre-assignment Details: Study consisted of 2 parts: Dose Escalation and Expansion. Enrollment of participants in Dose Expansion Part was planned to start after completion of Dose Escalation Part. Due to early termination of study, Dose Expansion Part was not conducted.
Groups:
- SAR440234: SAR440234 was administered as intravenous (IV) infusion once weekly for 6 weeks per Cycle. Per plan, participants were to receive first 2 to 3 doses as Lead-in doses followed by a fixed dose until the end of treatment or unless the dose needs to be decreased for safety reasons. Due to early study termination, all participants received only 1 treatment cycle at a dose of 1 nanogram per kilogram (ng/kg) once weekly.
Period: Overall Study
Arm/Group | SAR440234
Started | 7
Completed | 0
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Progressive disease | 5
Not completed — Sponsor's decision | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety population which included all registered participants who had given their informed consent and had received at least 1 dose of SAR440234.
Arm/Group | SAR440234
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation Part: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs: occurrence of any of following related to investigational medicinal product (IMP): Any grade (G) greater than or equal to (>=) 3 nonhematological adverse events (AE); G4 hematological toxicities (bone marrow hypocellularity, decreased neutrophils, febrile neutropenia, decreased platelet count and anemia) as defined in national cancer institute common terminology criteria for adverse events (NCI-CTCAE, v4.03); G3 or G4 cytokine release syndrome (CRS) (G1: fever, nausea, fatigue, headache, myalgias and malaise; G2: oxygen requirement less than [<] 40 percent (%); G3: oxygen requirement greater than [>] 40% ; G4: life-threatening symptoms, requirement for mechanical ventilation, organ toxicity, G5: death) graded by NCI Consensus Guidelines; Grade 2 CRS for >48 hours or <48 hours before IMP; any treatment-emergent AE of potential significance and IMP-related adverse reaction lasted >2 weeks with failure to recover to baseline or improve to Grade less than or equal to (<=1).
Time Frame: Cycle 1 (42 days)
Population: Analysis was performed on dose-limiting toxicities (DLT) evaluable population which included all participants in dose escalation part, who received at least 5 out of 6, weekly IV administrations of SAR440234 and participants who discontinued IMP before completion of Cycle 1 because of DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | SAR440234
Number analyzed (Participants) | 7
Participants | 1

2. Primary Outcome: Dose Escalation Part: Number of Participants With Allergic Reactions/Hypersensitivity and Cytokine Release Syndrome/Acute Infusion Reactions
Description: In this outcome measure, number of participants with allergic reactions or hypersensitivity and CRS or acute infusion reactions is reported. CRS is a nonantigen specific toxicity that occurs as result of potent immune activation mediated by large, rapid release of cytokines into blood from immune cells affected by IMP. Grading and management of CRS was based on National Cancer Institute (NCI) Consensus Guidelines 2014. Allergic/Hypersensitivity reactions or acute infusion reactions are defined as disorder characterized by adverse local/general response from exposure to allergen; graded by NCI CTCAE v4.03.
Time Frame: First IMP administration (Day 1) up to last dose of IMP + 30 days (i.e., up to 72 days)
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | SAR440234
Number analyzed (Participants) | 7
Participants | 2

3. Primary Outcome: Expansion Part: Percentage of Participants With Overall Response (OR) Per International Working Group (IWG) Criteria
Description: Response: assessed by IWG 2003 recommendations for acute myeloid leukemia (AML) and revised 2000 criteria for myelodysplastic syndrome (MDS). MDS - OR: complete remission (CR)/marrow CR/partial remission (PR), CR: repeat bone marrow show <5% myeloblasts and peripheral blood evaluations lasting >=2 months hemoglobin (>11 grams per deciliter), neutrophils 1500 per cubic millimeter (mm^3), platelets >=100000/mm^3, blasts 0% and no dysplasia, PR: all CR criteria except blasts decreased by >=50% over pretreatment or less advanced than pretreatment. AML - OR:CR/CR with incomplete hematological recovery(CRi)/PR, CR:absolute neutrophil count (ANC) >=1000 per microliter (mcL), platelets >=100000/mcL, <5% blast cells in bone marrow; auer rods should not be detectable; no platelet/whole blood transfusions for 7 days prior hematology test. CRi:all criteria of CR except platelets and/or ANC. PR:all CR criteria except blasts decreased by >=50% over pretreatment or less advanced than pretreatment.
Time Frame: From the date of first IMP administration until disease progression or death, whichever came earlier (up to 42 days)
Population: Due to the early termination of the study, data for this outcome measure was not collected and analyzed.
Arm/Group | SAR440234
Number analyzed (Participants) | 0

4. Primary Outcome: Expansion Part: Duration of Response (DOR)
Description: DOR: time from first tumor assessment at which the overall response was recorded as CR, marrow CR, or PR (MDS) and CR/CRi (AML) until documented progressive disease (PD) determined by IWG criteria, or death from any cause, whichever occurred first. Per IWG criteria, relapse was defined as reappearance of blasts in blood or bone marrow (>5%) or in any extramedullary site after a CR. CR:<= 5% myeloblasts in bone marrow with no evidence of persistent dysplasia; peripheral blood showing hemoglobin>=11g/dL. Marrow CR: no circulating blasts, <5% blast, absolute neutrophil count >1000/mcL, platelets >100000/mcL, no recurrence for 4 weeks. CRi: meet all criteria for CR except platelet count and/or ANC. PR: all CR criteria except blasts decreased by >=50% over pretreatment or less advanced than pretreatment. Progression: at least 50% decrease from maximum remission/response in granulocytes/platelets; reduction in Hgb by >=2 g/dL; transfusion dependence.
Time Frame: From 1st documentation of response to date of first documentation of disease progression or death, whichever came earlier (up to 42 days)
Population: Due to the early termination of the study, data for this outcome measure was not collected and analyzed.
Arm/Group | SAR440234
Number analyzed (Participants) | 0

5. Primary Outcome: Expansion Part: Number of Participants With Disease-free Survival
Description: Disease-free survival was defined as the time from date of first administration of study intervention until the earliest of any of the following: date of death or date of first response assessment confirming relapse or date of final response assessment which fails to confirm response whichever occurred first.
Time Frame: First IMP administration to date of first documentation of disease progression or relapse or death, whichever came earlier (up to 42 days)
Population: Due to the early termination of the study, data for this outcome measure was not collected and analyzed.
Arm/Group | SAR440234
Number analyzed (Participants) | 0

6. Secondary Outcome: Dose Escalation Part: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily had to have a causal relationship with the treatment. Serious AEs (SAEs) were any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. TEAEs were defined as the AEs that developed or worsened or became serious during the TEAE period (defined as the time from the first dose of the IMP to the last dose of IMP + 30 days).
Time Frame: From Baseline (Day 1) up to last dose of IMP + 30 days (i.e., up to 72 days)
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | SAR440234
Number analyzed (Participants) | 7
Participants
  Any TEAE | 7
  Any TESAE | 6

7. Secondary Outcome: Dose Escalation Part: Percentage of Participants With Objective Response Per IWG Criteria
Description: Objective response was defined as the percentage of participants who had a marrow CR, or PR (MDS) and CR/CRi (AML) per IWG criteria. For MDS, CR: repeat bone marrow show <5% myeloblasts and peripheral blood evaluations lasting >=2 months of hemoglobin (>11 g/dL), neutrophils 1500/mm^3, platelets >=100000/mm^3, blasts 0% and no dysplasia, PR: all CR criteria except blasts decreased by >=50% over pretreatment or less advanced than pretreatment. For AML, CR: ANC >=1000/mcL, platelet count >=100000/mcL, bone marrow should contain <5% blast cells; auer rods should not be detectable; no platelet/whole blood transfusions for 7 days prior to date of hematology assessment. CRi: morphologic complete remission but ANC count might be <1000/mcL or platelet <100000/mcL.
Time Frame: From the date of first IMP administration until disease progression or death, whichever came earlier (up to 42 days)
Population: Due to the early termination of the study, data for this outcome measure was not collected and analyzed.
Arm/Group | SAR440234
Number analyzed (Participants) | 0

8. Secondary Outcome: Immunogenicity: Number of Participants With Treatment-Emergent Anti-drug Antibodies (ADA) Response
Description: ADA response categories: 1) Treatment-induced ADA: Participants without pre-existing ADA and without pre-treatment samples and who developed ADAs during the TEAE period. 2) Treatment-boosted ADA: Participant with pre-existing ADAs that was increased at least a 4-fold in titer compared to Baseline during the TEAE period. 2) Treatment-emergent ADA: Participants with at least one treatment-induced/boosted ADA sample. TEAE period was defined as the time from the first dose of the IMP to the last dose of the IMP + 30 days.
Time Frame: From Baseline (Day 1) up to last dose of IMP + 30 days (i.e., up to 72 days)
Population: Analysis was performed on ADA population which included all participants who had given their informed consent, had received at least 1 dose (even incomplete) of SAR440234 and had at least 1 available ADA result after IMP administration.
Measure: Count of Participants; unit: Participants
Arm/Group | SAR440234
Number analyzed (Participants) | 7
Participants | 1

9. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Plasma Concentration (Cmax) of SAR440234
Description: Cmax was the maximum observed plasma concentration. Cmax was obtained by a non-compartmental analysis. Here in the time frame, Day = D, start of infusion = SOI, mid of infusion = MOI, end of infusion = EOI and hours = H.
Time Frame: Cycle 1: D 1: SOI, EOI, 1, 2, 5, 7, 24, 48, 72 H post EOI; D 8: SOI, MOI, EOI, 2, 5, 168 H post EOI; D 15: MOI, EOI, 2, 5, 24 H post EOI; D 22: SOI, MOI, EOI, 2, 5, 24, 48, 72, 96, 168 H post EOI; D 29: EOI, 2 H post EOI; D 36: SOI, EOI, 2 H post EOI
Population: Analyzed on PK population which included participants who had given their informed consent and had received at least one dose (even incomplete) of SAR440234 with at least 1 evaluable drug concentration after IMP administration. Here, number analyzed = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | SAR440234
Number analyzed (Participants) | 7
picograms per milliliter
  Cycle 1 Day 1 | 64.7 (171)
  Cycle 1 Day 8 | NA (NA) — Mean and standard deviation (SD) were not estimable as no participant had plasma concentration greater than lower limit of quantification.
  Cycle 1 Day 15: number analyzed (Participants) | 5
  Cycle 1 Day 15 | 99.1 (115)
  Cycle 1 Day 22: number analyzed (Participants) | 5
  Cycle 1 Day 22 | 57.1 (22.6)
  Cycle 1 Day 29: number analyzed (Participants) | 3
  Cycle 1 Day 29 | 74.5 (90.3)
  Cycle 1 Day 36: number analyzed (Participants) | 1
  Cycle 1 Day 36 | 70.4

ADVERSE EVENTS:
Time Frame: From first dose of IMP up to 30 days after the last dose of IMP (i.e., up to 72 days)
Description: Reported AEs and deaths were TEAEs that developed/worsened in grade or became serious during TEAE period (defined as the time from the first dose of the IMP to the last dose of IMP + 30 days). Analysis was performed on safety population.
Arm/Group | SAR440234
All-Cause Mortality (participants affected / at risk) | 2/7
Serious Adverse Events (participants affected / at risk) | 6/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAR440234 (N=7)
Alanine Aminotransferase Increased (Investigations) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Perirectal Abscess (Infections and infestations) | 1 (1)
Pneumonia Moraxella (Infections and infestations) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Cytokine Release Syndrome (Immune system disorders) | 1 (1)
Disease Progression (General disorders) | 3 (3)
Pyrexia (General disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAR440234 (N=7)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 2 (2)
Blood Alkaline Phosphatase Increased (Investigations) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (5)
Deafness (Ear and labyrinth disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Gingival Bleeding (Gastrointestinal disorders) | 1 (1)
Gingival Hypertrophy (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Oral Disorder (Gastrointestinal disorders) | 1 (2)
Proctalgia (Gastrointestinal disorders) | 1 (1)
Micturition Urgency (Renal and urinary disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Hypo Hdl Cholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2)
Oral Candidiasis (Infections and infestations) | 1 (1)
Staphylococcal Bacteraemia (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Cytokine Release Syndrome (Immune system disorders) | 2 (2)
Asthenia (General disorders) | 3 (3)
Chest Discomfort (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Gait Disturbance (General disorders) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (5)
Tenderness (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Sponsor decided to prioritize development of other novel therapies with more innovative mechanisms of action for R/R AML and other cancers. Thus, decided to terminate the study and stopped enrollment in Dose Expansion Part.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/55/NCT03594955/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT03594955/SAP_001.pdf